CLINICAL TRIAL: NCT06607432
Title: Use of Alpha-frequency Deep Transcranial Interference Stimulation (tIS) to Understand and Modify Temporal Dynamics of Face Emotion Recognition and Social/Affective Function
Brief Title: Temporal Interference Stimulation for Social Cognition
Acronym: TISSC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Daniel C. Javitt, MD, Professor of Psychiatry, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAV1631 (Stage 1a); 1U01MH135436 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy Controls
Keywords: Transcranial Interference Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The blind will be maintained by the Nathan Kline Institute (NKI) Data management group. Treatment assignment will be transmitted from the NKI Data management group directly to an unblinded research technician who will supervise the stimulation but will not otherwise perform ratings. The research technician will be instructed not to discuss treatment assignment with other members of the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active tIS 0.30 V/m and Sham (Active Comparator): Group 1 with 10 participants to receive a dose of 0.30 V/m and sham. The order of the intervention will be randomized.
  Interventions: Device: Transcranial Interference Stimulation (tIS); Other: Sham tIS
- Active tIS 0.35 V/m and Sham (Active Comparator): Group 2 with 10 participants to receive a dose of 0.35 V/m and sham. The order of the intervention will be randomized.
  Interventions: Device: Transcranial Interference Stimulation (tIS); Other: Sham tIS
- Active tIS 0.40 V/m and Sham (Active Comparator): Group 3 with 10 participants to receive a dose of 0.40 V/m and sham. The order of the intervention will be randomized.
  Interventions: Device: Transcranial Interference Stimulation (tIS); Other: Sham tIS

INTERVENTIONS:
Device: Transcranial Interference Stimulation (tIS) — Field strength dose of 0.30 - 0.40 V/m
  Other Names: Interference frequency stimulation (IFS); Transcranial Interference (TI)
Other: Sham tIS — Sham transcranial interferential stimulation. Sham comparator to be administered to all groups.

SUMMARY:
The long-term goal of this project is to evaluate whether a procedure termed transcranial interference stimulation (tIS) may be useful in the future in the treatment of severe neuropsychiatric disorders such as schizophrenia. The purpose of this stage of the project is to evaluate the safety and tolerability of tIS administration in healthy volunteers.

This study involves 30 healthy participants without known psychiatric illness, who will participate in groups of 10. The dose of tIS will be escalated progressively across doses. Functional magnetic resonance imaging (fMRI), magnetic resonance spectroscopy (MRS) and side effect checklists will be used to assess tIS safety/tolerability at each dose. In addition, electroencephalogram (EEG) will be collected simultaneously with tIS and used to assess target engagement. Face emotion recognition (FER) data will also be collected, but will be used for feasibility assessment only.

If successful, these studies will form the basis for future studies in schizophrenia.

DETAILED DESCRIPTION:
Transcranial interference stimulation (tIS) has been used outside of the United States (US) but not previously under Food and Drug Administration (FDA) regulation. This represents the first in human use of tIS in the US. tIS may be useful in the treatment of social cognitive impairments in schizophrenia and especially in the reversal of oscillatory dysfunction of the pulvinar nucleus of the thalamus. The overall project will investigate the safety and tolerability of tIS first in healthy volunteers and then in individuals with schizophrenia. This protocol is for stage 1a of the overall project only. In this stage, safety and tolerability will be assessed along with initial evaluation of target engagement. This stage uses a single ascending dose design with 10 participants per dose at each of three doses.

The stage 1a involves 30 healthy individuals and employs advanced techniques such as simultaneous electroencephalogram (EEG)/tIS, functional magnetic resonance imaging (fMRI), and magnetic resonance spectroscopy (MRS) to investigate the spatio-temporal dynamics of face emotion processing. These methods help us pinpoint specific brain regions like the pulvinar nucleus of the thalamus (PuN) and assess the safety and potential therapeutic benefits of tIS. Participants initially undergo an MRI session to localize their individual pulvinar nucleus of the thalamus (PuN). This step allows the investigators to model transcranial current flow accurately and precisely target the PuN using tIS. Subsequently, participants engage in simultaneous EEG recordings and tIS, which falls under the umbrella of transcranial electrical stimulation (tES). The timing of these sessions, whether single or repeated, depends on the study stage. The investigators also assess brain metabolism effects through MRS before and after tIS stimulation. Participants will go through several steps: 1) Interviews to determine eligibility 2) Behavioral tests of their ability to detect and interpret visual stimuli 3) "Brain wave" recordings or electroencephalogram 4) A non-invasive brain stimulation technique termed transcranial interference stimulation 5) Magnetic resonance imaging (MRI). Participants will also have an electrocardiogram and medical examination to evaluate their general health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-55 years
* Wechsler Adult Intelligence Scale (WAIS) intelligence quotient (IQ) >70
* Competent and willing to sign informed consent.
* Shall not have been prescribed any standing medications for treatment of a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) Axis I psychiatric disorders within 90 days of the study and shall not have been prescribed standing opioid analgesic, anticonvulsant, antidementia, antidepressant, antimigraine, antipsychotic, anxiolytic, bipolar agents, central nervous system agents, or sedative/hypnotics within 90 days of the study even if for a non-psychiatric indication. Intermittent use of sedative/hypnotic medications is permitted, but these agents shall not be used within 48 hours of the tIS administration.
* Healthy relative to age-dependent expectation as determined by medical history and physical examination within 90 days of enrollment.

Exclusion Criteria:

* Has a history of an illness, disease, condition injury, or disability which, in the opinion of the principal investigator (PI), may interfere with the completion of all study requirements per protocol, impact the quality of the data, or the validity of the study results.
* Contraindication to MRI (e.g. metal implants, claustrophobia, pregnancy)
* On the Columbia-Suicide Severity Rating Scale (C-SSRS) Screen Version-Recent, answers YES to Question 3 and NO to Question 6 (Moderate Risk) or answers YES to Question 4, 5, or 6 (High Risk).
* Presence or positive history of significant medical illnesses, including high blood pressure(defined as systolic blood pressure (SBP) >140 or diastolic blood pressure (DBP) >90, low blood pressure (SBP <100, DBP <60), orthostatic blood pressure as baseline (change in mean arterial pressure [1/3 systolic + 2/3 diastolic] of >20%), cardiac illness, or clinical significant abnormal electrocardiogram (EKG), as determined by the site physician
* Women of childbearing potential who, at enrollment or during the study:

  * have a positive urine pregnancy test or a self-reported pregnancy;
  * are heterosexually active without usage of a medically acceptable, highly effective contraceptive method* ( 1% pregnancy rate); or
  * are planning to become pregnant during the course of this study, as determined by the PI, are excluded from study participation. Examples include tubal ligation, vasectomized partner, intrauterine device (IUD) or intrauterine system (IUS), and longacting reversible contraceptives (LARC).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Pulvinar nucleus (PuN) activation levels | Once at baseline (day 1) and twice during each phase (day 8, day 15): 1x following active stimulation, 1x following sham stimulation in randomized order across participants
  Pulvinar nucleus (PuN) activation levels as determined by functional magnetic resonance imaging (fMRI, safety)
  These analyses assess the degree to which presentation of a stimulus designed to activate the pulvinar nucleus leads to an increase in local activation as reflected in the fMRI response. Units will be % increase in signal strength during stimulation vs. baseline.
Amplitude of 10-Hz visual Steady-State Response (ssVEP) | Twice during each phase (day 8, day 15): 1x during active stimulation, 1x during sham stimulation in randomized order across participants
  (Target engagement) This measure is obtained simultaneously with tIS and reflects the response of visual cortex to repetitive stimulation. Response is measured in microvolt-squared (uV2).

SECONDARY OUTCOMES:
Brunoni safety scale | Following each tIS session (day 8, 15)
  The Brunoni scale is a self-report scale for potential side effects following tIS, including headache, neck pain, scalp pain, tingling, itching, burning sensation, skin redness, sleepiness, trouble concentrating, acute mood change and "other"; Scores range from 1 (no discomfort) to 5 (severe discomfort). HIgher scores indicate greater severity.
Wong-Baker safety scale | Following each tIS session (day 8, 15)
  The Wong-Baker uses emotion faces to allow individuals to indicate the level of discomfort associated with the procedure. Scores range from 1 (no discomfort) to 5 (severe discomfort). Higher scores indicate greater discomfort.
Pulvinar nucleus (PuN) tissue levels of N-acetyl aspartate (NAA) | Once at baseline (day 1) and twice during each phase (day 8, 15): 1x following active stimulation, 1x following sham stimulation in randomized order across participants
  PuN tissue level of N-acetyl-aspartate (NAA)as determined by MRS (safety)
  NAA is a potential measure of oxidative stress. NAA levels will be measured as the amplitude of the NAA peak of the MRS spectrum.
Pulvinar nucleus (PuN) tissue levels of glutathione (GSH) | Once at baseline (day 1) and twice during each phase (day 8, 15): 1x following active stimulation, 1x following sham stimulation in randomized order across participants
  PuN tissue levels of glutathione (GSH), as determined by MRS (safety)
  GSH is a potential measure of oxidative stress. It will be defined based on the amplitude of the GSH peak in the MRS spectrum.
Columbia Suicide Severity Rating Scale (C-SSRS) | Days 1, 8, 15, 22
  The Columbia Suicide Severity Rating scale captures information on any thoughts you may be having regarding self-harm. The scale is scored from 0 (No thoughts) to 5 (Active suicidal ideation with plan and intent). Higher scores indicate more severe risk of suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Javitt, M.D., Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NewYork-Presbyterian Hospital (CUIMC/NYPH), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared via the NIMH Data Archives (NDA). Participants will be coded using global unique identifiers (GUIDs).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Sharing will be in accordance with NIMH Data Archive (NDA) policies and procedures (https://nda.nih.gov/)
Access Criteria: Data access will be in accordance with NIMH Data Archive (NDA) policies and procedures
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667